CLINICAL TRIAL: NCT06771869
Title: Sodium Balance Rather Than Fluid Balance as a Predictor of Respiratory Dysfunction in Critically Ill Septic Patients on Mechanical Ventilation; a Prospective Observational Study
Brief Title: Comparing Sodium to Fluid Balance in Predicting Respiratory Dysfunction in Critically Ill Septic Patients
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rania Maher Hussien, MD, Assistant professor, Ain Shams University
Other Study IDs: FMASU MS76/2024
Record Dates: First submitted 2025-01-08; First posted 2025-01-13 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Sodium Balance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Mechanically ventilated septic patients
  Interventions: Diagnostic Test: Sodium balance

INTERVENTIONS:
Diagnostic Test: Sodium balance — cumulative sodium balance and cumulative fluid balance will be estimated in the first three days after admission

SUMMARY:
Critically ill septic patients are at risk of positive sodium balance due to inadvertent excess administration, which may be over twice the daily requirement of sodium for healthy individuals This research will estimate sodium balance in critically ill septic patients on invasive mechanical ventilation (MV) for more than 48 hours and to evaluate the relationship between sodium balance and respiratory function (PaO2/FiO2 ratio) and length of MV

DETAILED DESCRIPTION:
This prospective observational cohort study assesses the effect of cumulative positive sodium balance on respiratory function in critically ill septic mechanically ventilated patients Patients admitted to the ICU for 6 months with Age more than 13 yrs. and less than 70 years, an APACHE II score of more than 12 is calculated on admission, and a SOFA score of more than 2 is calculated on admission. Septic patients who manifested by 2 or more of the following conditions: Temperature >38oC or <36oC, Heart rate >90 beats/min, Respiratory rate >20 breaths/min or PaCO2 <32mmHg, White blood cell count >12000/mm3, <4000/mm3 or >10% immature (band) forms, Mechanically ventilated patients for less than 48 hours and who were anticipated to be on MV for at least another 48 hours, Serum sodium concentration between 130 mmol/L and 150 mmol/L will be included in the study.

Data will be collected on the first three days after recruitment, with Day 1 being the day of enrollment. These include the Daily PaO2/FiO2 ratio, Daily urine output, and fluid balance. Routine laboratory investigations include Liver function tests, including ALT, AST, serum bilirubin, and serum albumin. Kidney function tests including serum creatinine and urea level. Complete blood count (CBC). Arterial blood gases. Serum lactate level.

Sodium and fluid intakes will be calculated and recorded for all solutions as the type and volume administered over each 24-hour study day for 3 days.

The primary outcome will be oxygenation (PaO2/FiO2 ratio) and length of MV stay while the Secondary outcomes include Length of ICU and hospital stay, ICU and hospital mortality, and SOFA scores at diagnosis of sepsis, Presence of shock (defined as requirement for vasopressor infusion at any dose for more than 6 hours).

* Labs specific for our study (on ICU admission and if needed):

  1. Procalcitonin (PCTQ).
  2. CRP.
* Serum electrolytes: Na, K, Ca

ELIGIBILITY:
Inclusion Criteria:

* APACHE II score of more than 12 calculated on admission.
* SOFA score of more than 2 calculated on admission.
* Septic patients who manifested by 2 or more of the following conditions:

  1. Temperature >38oC or <36oC
  2. Heart rate >90 beats/min
  3. Respiratory rate >20 breaths/min or PaCO2 <32mmHg.
  4. White blood cell count >12000/mm3, <4000/mm3 or >10% immature (band) forms.
* Mechanically ventilated patients for less than 48 hours and who were anticipated to be on MV for at least another 48 hours.
* Serum sodium concentration between 130 mmol/L and 150 mmol/L

Exclusion Criteria:

* Age less than 13 years and more than 70 years.
* Traumatic brain injury.
* ICU admission diagnosis of diabetic ketoacidosis, hyperosmolar hyperglycemic state, Child-Pugh class C liver cirrhosis, pregnancy or anticipated survival of less than 24 hours.
* Patients undergoing renal replacement therapy (RRT).

Ages: 13 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: mechanically ventilated septic patients
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
PaO2/FiO2 ratio | first three days after admission

SECONDARY OUTCOMES:
Length of ICU | first month after admission

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes